CLINICAL TRIAL: NCT02797587
Title: URBAN ARCH 4/5 Russia Cohort-Targeting HIV-comorbidities With Pharmacotherapy to Reduce Alcohol and Tobacco Use in HIV-infected Russians
Brief Title: Studying Partial-agonists for Ethanol and Tobacco Elimination in Russians With HIV (St PETER HIV)
Acronym: St PETER HIV
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Jeffrey Samet, Chief, Section of General and Internal Medicine, Boston Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: H-35288; U01AA020780 (NIH)
Record Dates: First submitted 2016-06-08; First posted 2016-06-13 (Estimated); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: HIV Infection; Alcohol Use; Smoking
Keywords: Alcohol Use; Tobacco Use; Smoking; Inflammation; Coronary Heart Disease; Russia; Varenicline; Cytisine; Nicotine Replacement Therapy; Partial Agonist Therapy; HIV; Reynolds risk score; VACS index
MeSH Terms: conditions — HIV Infections; Alcohol Drinking; Smoking; Tobacco Use; Inflammation; Coronary Disease | interventions — Varenicline; cytisine; Nicotine Replacement Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Varenicline + Nicotine Replacement Therapy placebo (Active Comparator): Study participants will receive active varenicline and be instructed to take the medication for 12 weeks; participants will also receive a placebo Nicotine Replacement Therapy mouth spray for 8 weeks.
  Interventions: Drug: Varenicline; Drug: Nicotine Replacement Therapy Placebo
- Varenicline placebo + Nicotine Replacement Therapy (Placebo Comparator): Study participants will receive placebo varenicline and be instructed to take the placebo medication for 12 weeks; participants will also receive an active Nicotine Replacement Therapy mouth spray for 8 weeks.
  Interventions: Drug: Nicotine Replacement Therapy; Drug: Varenicline Placebo
- Cytisine + Nicotine Replacement Therapy placebo (Active Comparator): Study participants will receive active cytisine and be instructed to take the medication for 25 days; participants will also receive a placebo Nicotine Replacement Therapy mouth spray for 8 weeks.
  Interventions: Drug: Cytisine; Drug: Nicotine Replacement Therapy Placebo
- Cytisine placebo + Nicotine Replacement Therapy (Placebo Comparator): Study participants will receive placebo cytisine and be instructed to take the medication for 25 days; participants will also receive an active Nicotine Replacement Therapy mouth spray for 8 weeks.
  Interventions: Drug: Nicotine Replacement Therapy; Drug: Cytisine Placebo

INTERVENTIONS:
Drug: Varenicline — 1 week starter kit followed by 1mg twice daily for 12 weeks.
  Arms: Varenicline + Nicotine Replacement Therapy placebo
Drug: Cytisine — Multi-daily dosing, range 3-9 mg daily for 25 days.
  Arms: Cytisine + Nicotine Replacement Therapy placebo
Drug: Nicotine Replacement Therapy — Mouth spray dosing based on standard recommendations tapered over 8 weeks.
  Arms: Cytisine placebo + Nicotine Replacement Therapy; Varenicline placebo + Nicotine Replacement Therapy
Drug: Varenicline Placebo — 1 week starter kit followed by 1 pill twice daily for 12 weeks.
  Arms: Varenicline placebo + Nicotine Replacement Therapy
Drug: Cytisine Placebo — Multi-daily dosing for 25 days.
  Arms: Cytisine placebo + Nicotine Replacement Therapy
Drug: Nicotine Replacement Therapy Placebo — Mouth spray dosing based on standard recommendations tapered over 8 weeks.
  Arms: Cytisine + Nicotine Replacement Therapy placebo; Varenicline + Nicotine Replacement Therapy placebo

SUMMARY:
This study is a randomized controlled trial (RCT) to compare the effects of varenicline, cytisine, and nicotine replacement therapy (NRT) to reduce: 1) alcohol use and craving, 2) smoking; and 3) inflammation and risk for coronary heart disease (CHD) and mortality among 400 HIV-infected Russians, with heavy alcohol consumption and tobacco use.

DETAILED DESCRIPTION:
HIV-infected heavy drinking smokers are at high risk for coronary heart disease (CHD) and death. The mechanisms driving increased CHD risk in HIV-infected people are unclear, but are linked to inflammation. HIV, heavy drinking, and smoking are all pro-inflammatory. HIV viral suppression with antiretroviral therapy does not eliminate the elevated CHD risk nor the increased inflammation (i.e., pre-HIV infection levels are not restored). Interventions that reduce alcohol use, smoking, or both in HIV-infected people could lower inflammation, CHD and death risk. Varenicline and cytisine are proven therapies for smoking cessation. When compared to placebo, varenicline has higher cessation rates than cytisine. Human trials suggest varenicline also has efficacy for reducing alcohol consumption and craving in heavy drinking smokers. In murine models, cytisine reduces alcohol consumption. The comparative efficacy of varenicline and cytisine to reduce alcohol consumption and by extension, inflammation, CHD, and mortality risk, in humans has not been tested, nor has their comparative effectiveness been tested for smoking. Neither drug has been tested for smoking cessation against nicotine replacement therapy (NRT) in HIV-infected heavy drinking smokers. Three compelling reasons to test varenicline and cytisine in HIV-infected heavy drinking smokers are: 1) both show promise in HIV-uninfected people; 2) the morbidity caused by heavy drinking and smoking in HIV-infected persons is significant; and 3) treating heavy drinking and smoking with one medication represents a significant advance in reducing polypharmacy and improving patient care. Thus, investigators propose a 4-arm placebo-controlled randomized controlled trial (RCT) among 400 HIV-infected heavy drinking smokers. Trial arms are varenicline+NRT placebo, cytisine+NRT placebo, NRT+varenicline placebo, NRT+cytisine placebo. All participants will receive counseling (alcohol & tobacco) and medications (placebo & active). Specific aims will compare effects of varenicline, cytisine, and NRT at 3 months on past month % heavy drinking days and alcohol craving, cigarettes per day and smoking abstinence (verified by carbon monoxide), inflammation (hsCRP, IL-6), CHD (Reynolds risk score), and mortality (VACS index) risk. Investigators hypothesize that (1) Varenicline has greater efficacy than NRT for reducing heavy drinking, smoking, inflammation, CHD and mortality risk; (2) Cytisine has greater efficacy than NRT; and (3) Varenicline has greater efficacy than cytisine for these outcomes. Investigators will conduct an RCT, Studying Partial-agonists for Ethanol and Tobacco Elimination in Russians with HIV (St PETER HIV), in a country with an HIV epidemic and high per-capita alcohol consumption and smoking. Investigators will recruit from the ongoing Russia ARCH cohort in St. Petersburg (part of our NIAAA funded HIV/AIDS Alcohol Consortium - URBAN ARCH). If investigator hypotheses are correct, St PETER HIV could make nicotinic partial-agonists standard care for HIV+ heavy drinking smokers, and lead to reduced inflammation, CHD and mortality risk through this "one drug, two diseases" approach. This trial addresses the paucity of RCT data to guide treatment of these CHD risk factors in HIV-infected people.

The Russia ARCH Cohort and the St PETER HIV study will draw from an established cohort of HIV-infected smokers and heavy drinkers to compare the effects of two partial nicotinic receptors, varenicline and cytisine, on alcohol consumption, alcohol craving, smoking, inflammation, CHD risk and mortality risk. St PETER HIV further addresses the paucity of randomized controlled trial data to guide treatment of heavy alcohol consumption and smoking in HIV-infected people.

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years old
* HIV-infected
* ≥ 5 heavy drinking days in the past 30 days (NIAAA at-risk drinking levels)
* Smoking an average of at least 5 cigarettes per day
* Provision of contact information for 2 contacts to assist with follow-up
* Stable address within 100 kilometers
* Possession of a telephone (home or cell)
* Interest in cutting down/quitting alcohol or tobacco
* Able and willing to comply with all study protocols and procedures

Exclusion Criteria:

* Not fluent in Russian
* Cognitive impairment
* Pregnant or planning to become pregnant in next 3 months
* Breastfeeding
* Unstable psychiatric illness (i.e. ,answered yes to any of the following: past three month a) active hallucinations; b) mental health symptoms prompting a visit to the ED or hospital; mental health medication changes due to worsening symptoms; presence of suicidal ideations)
* History of pheochromocytoma
* Taking smoking cessation medications in past 30 days
* History of seizures
* History of Buerger's disease
* Acute coronary syndrome within 1 month of enrollment
* Systolic BP > 180 mm Hg or diastolic BP > 105 mm Hg
* Currently taking anti-tuberculosis medications
* Currently taking Galantamine or Physostigmine
* BAC level of 0.10% or higher
* Known allergy to varenicline (Chantix) or cytisine (Tabex)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2017-07-19 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-12-15 (Actual)

PRIMARY OUTCOMES:
Percent heavy drinking days in past 30 days | Participants will be followed for up to 12 months (primary endpoint at 3 month)
  Self-reported past 30-day alcohol consumption obtained via the Timeline Followback (TLFB) method, heavy drinking defined by NIAAA definition

SECONDARY OUTCOMES:
Alcohol craving | Participants will be followed for up to 12 months (primary endpoint at 3 month)
  Measured by the Penn Alcohol Craving Scale
Carbon monoxide-validated smoking cessation | Participants will be followed for up to 12 months (primary endpoint at 3 month)
  Self-reported 7-day point prevalence abstinence and a carbon monoxide measured in end-expired air threshold of <10 ppm.
Coronary heart disease risk | Participants will be followed for up to 12 months (primary endpoint at 3 month)
  Measured by the Reynolds risk score
Mortality risk | Participants will be followed for up to 12 months (primary endpoint at 3 month)
  Measured by the VACS index
Cigarettes per day in past 7 days | Participants will be followed for up to 12 months (primary endpoint at 3 month)
  Self-report, obtained via Timeline Followback (TLFB) method
hsCRP levels | Participants will be followed for up to 12 months (primary endpoint at 3 month)
  Biomarker of inflammation measured via study test
IL-6 levels | Participants will be followed for up to 12 months (primary endpoint at 3 month)
  Biomarker of inflammation measured via study test

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey H Samet, MA, MA, MPH, Principal Investigator — Boston University/Boston Medical Center
Locations (1):
- First St. Petersburg Pavlov State Medical University, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: Yes
All data from the study will be placed into the URBAN ARCH repository.

REFERENCES:
- [Derived] Tindle HA, Freiberg MS, Cheng DM, Gnatienko N, Blokhina E, Yaroslavtseva T, Bendiks S, Patts G, Hahn J, So-Armah K, Stein MD, Bryant K, Lioznov D, Krupitsky E, Samet JH. Effectiveness of Varenicline and Cytisine for Alcohol Use Reduction Among People With HIV and Substance Use: A Randomized Clinical Trial. JAMA Netw Open. 2022 Aug 1;5(8):e2225129. doi: 10.1001/jamanetworkopen.2022.25129. PMID 35930287
- See also: URBAN ARCH, a member of NIAAA CHAART (Consortiums for HIV/AIDS & Alcohol Research Translation) initiative, conducts and disseminates interdisciplinary research on how alcohol impacts people with HIV and develops interventions to reduce related outcomes. — http://www.urbanarch.org